CLINICAL TRIAL: NCT06004388
Title: A Randomized, Double-Blind, Parallel-Group, Virtual Study to Evaluate the Efficacy and Safety of Two Prescription Digital Therapeutics for the Prevention of Episodic Migraine in Late Adolescents and Adults Currently Receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy
Brief Title: Study of Two Digital Therapeutics for the Prevention of Episodic Migraine Receiving CGRP Therapy (ReMMiD-C)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Click Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-132-R-002
Record Dates: First submitted 2023-07-26; First posted 2023-08-22 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-03

CONDITIONS: Migraine; Episodic Migraine; Headache; Headache, Migraine
Keywords: Prescription digital therapeutic (PDT); Software as a Medical Device (SaMD); Smartphone app; CGRP; Calcitonin Gene-Related Peptide Inhibitor Therapy
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- ReMMiD-C Therapeutic Arm A (Experimental): Mobile application A (ReMMiD-C Digital Therapeutic) as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy.
  Interventions: Device: Click Digital Therapeutic
- ReMMiD-C Therapeutic Arm B (Experimental): Mobile application B as a software-based intervention for the preventive treatment of episodic migraine in late adolescents and adults receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy.
  Interventions: Device: Click Digital Therapeutic

INTERVENTIONS:
Device: Click Digital Therapeutic — Evaluate the efficacy and safety of prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adults and adolescents receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy

SUMMARY:
Randomized study of two digital therapeutics for the prevention of episodic migraine in patients currently receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy

DETAILED DESCRIPTION:
The purpose of this randomized trial is to evaluate the efficacy and safety of two prescription mobile applications that provide an interactive, software-based intervention for the preventative treatment of episodic migraine in late adolescents and adults who are receiving Calcitonin Gene-Related Peptide (CGRP) Inhibitor Therapy.

ELIGIBILITY:
Inclusion Criteria:

* A participant will be eligible for entry into the study if all of the following criteria are met per participant self-report:
* Willing and able to provide written informed consent to participate in the study, attend study visits, and comply with study-related requirements and assessments.
* Lives in the United States.
* Adult or late adolescent, ≥ 18 years of age at the time of informed consent.
* Able to read and understand the English informed consent form.
* The following will be investigator-reviewed: Participant has at least a 1-year history of migraine (with or without aura) consistent with a diagnosis according to the International Classification of Headache Disorders (ICHD), 3rd Edition:

  i. Age of onset of migraines prior to 50 years of age

ii. Migraine attacks, on average, lasting 4-72 hours if untreated

iii. Per participant report, 4 or more migraine days per month within the last 3 months prior to the Screening Visit (a month is defined as 28 days)

iv. Four to fourteen migraine days during the run-in period

* Is currently managing migraines with at least 1 prescription CGRP inhibitor therapy for the preventive or acute treatment of episodic or chronic migraine during the 3 months prior to screening.
* Is the sole user of an iPhone with an iPhone operating system (iOS) 14 or later or a smartphone with an Android operating system (OS) 11 or later, and is willing to download and use the specified eDiary and Study App required by the protocol.
* Is willing and able to receive SMS text messages and push messages on their smartphone.
* Is the owner of, and has regular access to, an email address.
* Has regular access to the Internet via cellular data plan and/or wifi.
* Understands the use of and interest in the eDiary and the Study App during the screening period and the baseline visit (Day 1).

Exclusion Criteria:

* A participant will not be eligible for study entry if any of the following criteria are met per participant self-report:
* History of basilar migraine or hemiplegic migraine.
* Active chronic pain syndromes, such as fibromyalgia, chronic pelvic pain, or complex regional pain syndrome (CRPS).
* Other pain syndromes (including trigeminal neuralgia), psychiatric conditions (such as current major depressive episode, bipolar disorder, major depressive disorder, schizophrenia), dementia, or significant neurological disorders (other than migraine) that, in the Investigator's opinion, might interfere with study assessments.
* History of, treatment for, or evidence of, alcohol or drug abuse within the past 12 months (48 weeks) or having met DSM-5 criteria for any significant substance use disorder within the past 12 months (48 weeks) from the date of the screening visit.
* History of use of analgesics (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs] or acetaminophen, including opioids) or butalbital on ≥ 15 days per month during the 3 months (12 weeks) prior to the Screening Visit or during the run-in period.
* Post-traumatic headache, persistent post-traumatic headache, or post-concussion syndrome.
* Other significant acute or chronic medical condition(s) that, in the opinion of the Investigator, may confound the interpretation of findings to inform PDT development.
* Failure to adhere with or inability to complete eDiary inputs and onboarding activities during the run-in period. Participants who are not adherent during the run-in period are not eligible for study entry.
* Previous enrollment in any digital therapeutics pilot or pivotal study for a migraine indication.
* Participation in any other investigational clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-06-05 (Actual)

PRIMARY OUTCOMES:
Change in Monthly Migraine Days (MMDs) | Baseline to Week 12
  Change from baseline in the number of Monthly Migraine Days (MMDs) at Week 12

SECONDARY OUTCOMES:
Proportion of Patients with Decrease in MMDs | Baseline to Week 12
  Proportion of participants who have at least a 50% reduction from baseline in the mean number of MMDs at Week 12
Change in MMDs at Weeks 4 and 8 | Baseline to Weeks 4 and 8
  Change from baseline in the number of MMDs recorded over the previous 28 days at Week 4 and Week 8
Change in Mean MMDs | Baseline to Week 12
  Reduction from baseline in the mean number of MMDs over 12 weeks
Change in Average Headache Severity | Run-in to Weeks 9-12
  Change in the average severity of headache from the run-in period to Weeks 9-12
Change in Migraine Questionnaire | Baseline to Weeks 4, 8 and 12
  Change from baseline in the Migraine-Specific Quality-of-Life Questionnaire v2.1 (MSQ) at Week 4, Week 8, and Week 12
Change in Migraine Disability Assessment (MIDAS) | Baseline to Weeks 4, 8, and 12
  Change from baseline in the Migraine Disability Assessment (MIDAS) at Week 4, Week 8, and Week 12
Change in Migraine Medication Use (frequency) | Run-in to Weeks 9-12
  Change in the use (frequency) of acute migraine medications from the run-in period to Weeks 9-12
Change in Migraine Medication Use (dose) | Run-in to Weeks 9-12
  Change in the use (dose) of acute migraine medications from the run-in period to Weeks 9-12
Change in Migraine Medication Use (medication type) | Run-in to Weeks 9-12
  Change in the use (type) of acute migraine medications from the run-in period to Weeks 9-12

CONTACTS AND LOCATIONS:
Overall Officials: Shaheen Lakhan, Study Director — Click Therapeutics
Locations (1):
- Click Therapeutics, New York, New York, United States